CLINICAL TRIAL: NCT02125513
Title: Randomized Phase II Study of 3 vs 6 Courses of Neoadjuvant Carboplatin-paclitaxel Chemotherapy in Stage IIIC or IV Epithelial Ovarian Cancer, Fallopian Tube Carcinoma or Primary Peritoneal Carcinoma
Brief Title: Neoadjuvant Chemotherapy in Epithelial Ovarian Cancer
Acronym: GOGER-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Claudio Zamagni MD, MD Medical Oncologist, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOGER-01; 2013-002520-17 (EudraCT Number)
Record Dates: First submitted 2014-04-17; First posted 2014-04-29 (Estimated); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Carcinoma; Peritoneal Carcinoma
Keywords: neoadjuvant chemotherapy; ovarian cancer; fallopian tube carcinoma; peritoneal carcinoma; randomized study
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: 3 courses (Active Comparator): Patients will receive 3 courses of i.v. carboplatin AUC 5 and paclitaxel 175 mg/m2 every 3 weeks, followed by cytoreductive surgery within 6 weeks from the last cycle of chemotherapy. Alternatively, the Participating Centres can use the weekly paclitaxel schedule: carboplatin AUC 6 day 1 and paclitaxel 80 mg/m2 day 1-8-15.
  Interventions: Drug: carboplatin and paclitaxel followed by surgery
- Arm B: 6 courses (Experimental): Patients will receive 6 courses of i.v. carboplatin AUC 5 and paclitaxel 175 mg/m2 every 3 weeks, followed by cytoreductive surgery within 6 weeks from the last cycle of chemotherapy. Alternatively, the Participating Centres can use the weekly paclitaxel schedule: carboplatin AUC 6 day 1 and paclitaxel 80 mg/m2 day 1-8-15.
  Interventions: Drug: carboplatin and paclitaxel followed by surgery

INTERVENTIONS:
Drug: carboplatin and paclitaxel followed by surgery

SUMMARY:
The purpose of this study is to define whether 6 courses of neoadjuvant chemotherapy can lead to a higher rate of complete cytoreductive surgery compared with 3 courses of neoadjuvant chemotherapy in patients with epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years.
* Karnofsky Performance Scale ≥ 60%
* Histologically confirmed epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma with the exception of mucinous, clear cell, low-grade carcinoma and carcinosarcoma histologies.
* Documented International Federation of Gynecologic Oncology (FIGO) stage IIIC-IV oligometastatic unsuitable for complete primary cytoreductive surgery. Inoperability must be confirmed by open laparoscopy or by laparotomy.
* Adequate bone marrow, liver and renal function to receive chemotherapy and subsequently to undergo surgery:

  * white blood cells >3,000/µL, absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL, hemoglobin ≥9 g/dL,
  * serum creatinine <1.25 x upper normal limit (UNL) or creatinine clearance ≥60 mL/min according to Cockroft-Gault formula or to local lab measurement
  * serum bilirubin <1.25 x UNL, AST(SGOT) and ALT(SGPT) <2.5 x UNL.
* Signed informed consent obtained prior to any study-specific procedures

Exclusion Criteria:

* Mucinous, clear cell, low-grade carcinoma and carcinosarcoma histologies.
* Synchronous or previous other malignancies within 3 years prior to starting study treatment, with the exception of adequately treated non-melanomatous skin cancer or carcinoma in situ (of the cervix or breast or other sites).
* Patients with brain metastases, seizure not controlled with standard medical therapy, or history of cerebrovascular accident (CVA, stroke) or transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months from the enrollment on this study.
* Any other concurrent medical conditions contraindicating surgery or chemotherapy that could compromise the adherence to the protocol (including but not limited to impaired cardiac function or clinically significant cardiac diseases, active or uncontrolled infections, HIV-positive patients on antiretroviral therapy, uncontrolled diabetes, cirrhosis, chronic active or persistent hepatitis, impaired respiratory function requiring oxygen-dependence,serious psychiatric disorders).
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who obtain a complete cytoreduction (no macroscopic residual tumor) at surgery , as a comparative outcome measure of 3 vs 6 courses of neoadjuvant chemotherapy | within 6 weeks after the last cycle of chemotherapy
  The primary objective of this study is to define whether 6 courses of neoadjuvant chemotherapy can lead to a higher rate of complete cytoreductive surgery compared with 3 courses of neoadjuvant chemotherapy in patients with bulky stage IIIC or IV epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer

SECONDARY OUTCOMES:
Percentage of patients with grade 3-5 perioperative toxicity (according to CTCAE), as a measure of safety | within 30 days after surgery
  To determine whether a longer duration of neoadjuvant chemotherapy is associated with a lower rate of perioperative grade 3-5 toxicities. The surgical adverse events are defined as:
  * intraoperative, which occur during surgical procedure
  * perioperative , which occur from day 1 to day 7 after surgery
  * postoperative, which occur from day 8 to 30 days after surgery
  Adverse events list for surgical procedures:
  Postoperative death (<30 days); Hemorrhage/bleeding intraoperative or postoperative requiring at least transfusion of 2 units of non-autologous red blood cells; Vascular events: thrombosis/embolism, disabling or life-threatening vessel injury-artery or vein, symptomatic or life-threatening visceral arterial ischemia; Infections requiring IV antibiotics, antifungal or antiviral interventions or at risk for life-threatening consequences; Gastrointestinal fistula; Urinary fistula; Lymphocele, requiring medical or operative intervention.
Percentage of patients with pathological complete response | after surgery, up to 1 month after surgery
  To determine whether a longer duration of neoadjuvant chemotherapy is associated with higher rate of pathological complete response.
  Complete pathological response is defined as the absence of cancer cells in surgical specimens, and very good partial remission is defined as the persistence of only small clusters (< 1 cm) or individual cancer cells and no macroscopic residual after surgery. Partial pathological remission is defined as a tumor burden reduction between 30 and 90% at surgery, while stable disease is defined as no tumour burden reduction or reduction lower than 30% at surgery, compared with initial diagnostic laparoscopy. Only patients with complete and very good partial remissions are considered as pathological responders, while all the other cases are considered as pathological non-responders.
Rate of progression-free survival | from date of randomization until the date of disease progression or second cancer or death from any cause, whichever occurs first, assessed for 10 years after the end of chemotherapy
  To determine whether a longer duration of neoadjuvant chemotherapy is associated with longer progression-free survival.
Health related quality of life | from baseline to safety follow-up visit (30-34 days after surgery)
  To compare the quality of life in the two treatment groups
Rate of radiological responses | at the end of neoadjuvant chemotherapy, before surgery
  To determine whether a longer duration of neoadjuvant chemotherapy is associated with a higher rate of radiological responses (according to RECIST 1.1 criteria).
Rate of decrease of CA125 levels during NACT | from cycle 1 of chemotherapy to safety follow-up visit (30-34 days after surgery)
  To determine whether a longer duration of neoadjuvant chemotherapy is associated with a greater decrease of CA125 levels.
Rate of overall survival | from date of randomization until date of death due to any cause, assessed until 10 years after the end of chemotherapy
  To determine whether a longer duration of neoadjuvant chemotherapy is associated with longer overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Zamagni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (5):
- Italy (5):
  - S.Orsola-Malpighi Hospital, Bologna
  - Azienda Ospedaliero-Universitaria di Parma - Oncologia Medica, Parma
  - IRCCS Ospedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario A. Gemelli, Rome
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia di Udine, Reparto di Oncologia, Udine